CLINICAL TRIAL: NCT07051278
Title: ABL90 FLEX PLUS Method Comparison Study for ctBil and FHbF in Neonatal Capillary Whole Blood
Brief Title: ABL90 FLEX PLUS Method Comparison Neonatal Capillary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radiometer Medical ApS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DC-083186
Record Dates: First submitted 2024-05-30; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Method Comparison for ABL90 FLEX PLUS in Neonatal Subjects
Keywords: Blood Gas; Method Comparison; Capillary; Neonates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Investigational Device (Active Comparator): The Investigational Device in this clinical study is the ABL90 FLEX PLUS running SW3.5 MR2 manufactured by Radiometer Medical ApS. The analyzer provides results for 17 parameters in 35 seconds using 65 μL heparinized whole blood. However, in this investigation only the data concerning the parameters ctBil and FHbF will be evaluated.
  Interventions: Device: Method Comparison
- Predicate device (Sham Comparator): The predicate device for this study is the unmodified device ABL90 FLEX PLUS (k160153) running software SW 3.1 MR7 including sensor casettes and solution packs versions corresponding to 2016.
  ABL90 FLEX PLUS SW 3.1 MR7, has been selected as the predicate device because it has the appropriate 510(k) clearance, and the intended use matches the ABL90 FLEX PLUS SW. SW3.5 MR2 device.
  Interventions: Device: Method Comparison

INTERVENTIONS:
Device: Method Comparison — Quantifying the relationship using comparison measurement from the same sample between ABL90 FLEX PLUS and the predicate device within the reportable range for ctBil and FHbF in heparinized capillary whole blood samples in capillary measuring mode (C65).

SUMMARY:
The study is intended to validate performance claims for method comparison for ABL90 FLEX PLUS in heparinized neonatal capillary whole blood for ctBil and FHbF in a POC setting

DETAILED DESCRIPTION:
The objective is to perform a method comparison study to quantify the relationship using comparison measurement from the same sample between ABL90 FLEX PLUS and the predicate device within the reportable range for ctBil and FHbF in heparinized capillary whole blood samples in capillary measuring mode (C65).

This study will together with a method comparison study performed with surrogate capillary samples contribute to the overall validation of the performance of ABL90 FLEX for capillary whole blood with regards to the parameters ctBil and FHbF measured using the capillary mode.

This study is anticipated to run for approximately 6-12 months from site initiation visit till close-out visit depending on patient enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent collected from legal representative able to understand information given and willing and able to voluntary give their consent to participate in this study.
* The age of the subject must be ≤28 days.
* Subject evaluated as suitable according to the protocol to enrol in the study by principal investigator or designee

Exclusion Criteria:

* Subject where sample collection is evaluated by principal investigator or designee to impose an unnecessary risk.
* Subject, who has an invalid written informed consent or has withdrawn consent.
* Subject who has already provided successful results from capillary samples, to cover both parameters.
* Subjects exposed to the substances listed in Appendix 1 with last dose within 72 hours, should be excluded due to risk of interference.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 129 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Primary Endpoints | 12 months
  Bias between device under investigation and comparative device at medical decision level across sites; (unit is mg/dL)

SECONDARY OUTCOMES:
Secondary Endpoints | 12 months
  Bias between device under investigation and comparative device at a medical decision point in native capillary samples per site; (unit is mg/dL)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Albert Einstein College of Medicine, The Bronx, New York
  - Duke University, Durham, North Carolina
  - University of Virginia, Charlottesville, Virginia